CLINICAL TRIAL: NCT00871546
Title: A Randomized Phase 2 Study of SCH 727965 in Subjects With Relapsed or Refractory Mantle Cell Lymphoma (MCL) or B-Cell Chronic Lymphocytic Leukemia (B-CLL)
Brief Title: SCH 727965 in Patients With Mantle Cell Lymphoma or B-Cell Chronic Lymphocytic Leukemia (Study P04715)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P04715
Record Dates: First submitted 2009-03-26; First posted 2009-03-30 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-08

CONDITIONS: Lymphoma, Mantle-Cell; Leukemia, Lymphocytic, Chronic, B-Cell
MeSH Terms: conditions — Lymphoma, Mantle-Cell; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — dinaciclib; Bortezomib; Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Participants with MCL randomized to SCH 727965 (Experimental)
  Interventions: Drug: SCH 727965
- Participants with MCL randomized to bortezomib (Active Comparator)
  Interventions: Drug: Bortezomib
- MCL treated w/SCH 727965 after progression on bortezomib (Experimental)
  Interventions: Drug: SCH 727965
- Participants with B-CLL randomized to SCH 727965 (Experimental)
  Interventions: Drug: SCH 727965
- Participants with B-CLL randomized to alemtuzumab (Active Comparator)
  Interventions: Biological: Alemtuzumab
- B-CLL treated w/ SCH 727965 after progression on alemtuzumab (Experimental)
  Interventions: Drug: SCH 727965

INTERVENTIONS:
Drug: SCH 727965 — SCH 727965 50 mg/m2 IV on Day 1 of each 21-day cycle until disease progression.
  Arms: B-CLL treated w/ SCH 727965 after progression on alemtuzumab; MCL treated w/SCH 727965 after progression on bortezomib; Participants with B-CLL randomized to SCH 727965; Participants with MCL randomized to SCH 727965
Drug: Bortezomib — Bortezomib 1.3 mg/m2 IV on Days 1, 4, 8, and 11 of each 21-day cycle until disease progression.
  Other Names: Velcade
  Arms: Participants with MCL randomized to bortezomib
Biological: Alemtuzumab — Alemtuzumab dose-titrated to the goal maintenance dose of 30 mg/day IV or SC three times a week on alternate days for a total of 12 weeks.
  Other Names: Campath
  Arms: Participants with B-CLL randomized to alemtuzumab

SUMMARY:
Participants will be randomized to SCH 727965 or a comparator drug (bortezomib for mantle cell lymphoma [MCL] or alemtuzumab for B cell chronic lymphocytic leukemia [B CLL]). Part 1 of the study will determine the activity of SCH 727965 treatment in participants with MCL and participants with B-CLL. Part 2 of the study will determine the activity of SCH 727965 treatment in participants who experienced disease progression after standard treatment with the comparator drug during Part 1.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 years, either sex, any race.
* Eastern Cooperative Oncology group performance status of 0 or 1.
* Adequate hematologic, renal, and hepatic organ function and laboratory parameters.
* For subjects with MCL:

  * Diagnosis of MCL according to the World Health Organization (WHO) criteria.
  * Received at least one prior chemotherapeutic regimen, but no more than two regimens including stem cell transplantation..
  * Measurable or assessable disease by the Revised Response Criteria for Malignant Lymphoma.
* For subjects with B-CLL

  * Documented B-CLL according to the National Cancer Institute Working Group (NCI-WG) criteria.
  * Received at least one prior alkylating agent-based regimen and one fludarabine- or pentostatin-containing regimen, but must not have received more than two prior regimens.
  * Measurable or assessable disease by NCI-WG criteria.

Exclusion Criteria:

* Known central nervous system involvement of MCL or B-CLL.
* Previous treatment with SCH 727965 or other cyclin-dependent kinase inhibitors.
* For MCL, previous treatment with bortezomib.
* For B-CLL, previous treatment with alemtuzumab.
* Known HIV infection.
* Known active hepatitis B or C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2009-03; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Response rate of initial treatment with SCH 727965 in subjects with MCL or B-CLL. | Time to identified disease progression on SCH 727965 in Part 1 (approx. 6 months)
Response rate in subjects treated with SCH 727965 after disease progression on comparator drug. | Time to identified disease progression on SCH 727965 in Part 2 (approx. 6 months)

SECONDARY OUTCOMES:
Time to disease progression for initial treatment with SCH 727965. | Time to identified disease progression on SCH 727965 in Part 1 (approx. 6 months)
Time to disease progression and response rate for treatment with the comparator drug. | Time to identified disease progression on comparator drug (bortezomib for MCL or alemtuzumab for B-CLL).
Response rate for treatment with the comparator drug. | Time to identified disease progression on comparator drug (bortezomib for MCL or alemtuzumab for B-CLL).
Time to disease progression in participants treated with SCH 727965 after disease progression on comparator drug. | Time to identified disease progression on SCH 727965 in Part 2 (approx. 6 months)